CLINICAL TRIAL: NCT07323784
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Efficacy of NTX-1472, a V1a Receptor Antagonist, in Adults With Social Anxiety Disorder
Brief Title: A Study of NTX-1472 in Social Anxiety Disorder
Acronym: SOAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Newleos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTX-1472-201
Record Dates: First submitted 2026-01-06; First posted 2026-01-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety Disorder (SAD)
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NTX-1472 (Experimental)
  Interventions: Drug: NTX-1472
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTX-1472 — Daily (QD) x 8 weeks.
  Arms: NTX-1472
Drug: Placebo — Daily (QD) x 8 weeks.
  Arms: Placebo

SUMMARY:
The primary goal of this Phase 2 clinical trial is to determine the effects of a novel V1a receptor antagonist (NTX-1472) in adults with Social Anxiety Disorder (SAD). The main questions this trial aims to answer are:

* Is NTX-1472 safe and well tolerated in adults with SAD?
* How effectively does NTX-1472 treat adults with SAD?

Researchers will compare the effects of NTX-1472 with matching placebo (a look-alike capsule that contains no drug).

Participants will:

* Take NTX-1472 or matching placebo every day for 8 weeks
* Visit the clinic 6 times over the course of 14 weeks for checkups and tests

ELIGIBILITY:
Key Inclusion Criteria

* Has provided written informed consent for the study and is willing to comply with all requirements of the protocol
* English speaker
* Male or female, ≥18 and ≤65 years of age
* Current diagnosis of generalized Social Anxiety Disorder (SAD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) and confirmed by the Structured Clinical Interview for DSM-5 (SCID-5-CT).
* Clinician-administered Liebowitz Social Anxiety Score (LSAS) total score ≥70 at Screening
* Clinician-rated Hamilton Depression Rating Scale (HDRS 17) (17 items) total score <16 at Screening
* If participant is of childbearing potential, must commit to practicing effective methods of birth control during the study and at least 14 days after the last dose.

Key Exclusion Criteria

* Current diagnosis of performance-only SAD as defined by the DSM-5 and confirmed by the SCID-5-CT.
* Current diagnosis of any of the following psychiatric condition(s) as defined by the DSM-5 (participants with current generalized anxiety disorder may be included): Attention-deficit/hyperactivity disorder, Autism spectrum disorder, Major depressive disorder, Personality disorder, Post-traumatic stress disorder.
* Past or current diagnosis of any of the following psychiatric condition(s), as defined by the DSM-5: Bipolar disorder, Feeding and eating disorder (in adulthood), Obsessive-compulsive disorder, Schizophrenia spectrum or other psychotic disorder, Substance use disorder (within 12 months of Screening).
* Receiving daily psychotropics within 4 weeks of Screening
* Is at risk for suicidal ideation as per C-SSRS
* Has moderate or severe hepatic impairment
* Has severe renal impairment
* Women who are pregnant or women who are currently breastfeeding unless they are willing to stop breastfeeding for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Baseline to Week 8

SECONDARY OUTCOMES:
Change in the clinician-administered Liebowitz Social Anxiety Scale (LSAS) total score | Baseline to Week 8
  The Liebowitz Social Anxiety Scale (LSAS) is a clinician-administered scale that is designed to record the severity of subjective anxiety and avoidance behavior across a range of social interaction and performance situations. The fear and avoidance subscale scores range from 0 to 72 each. The total score ranges from 0 to 144. Higher scores indicate greater severity of social anxiety.
Change in LSAS Fear/Anxiety and Avoidance subscale score | Baseline to Week 8
  The Liebowitz Social Anxiety Scale (LSAS) is a clinician-administered scale that is designed to record the severity of subjective anxiety and avoidance behavior across a range of social interaction and performance situations. The fear and avoidance subscale scores range from 0 to 72 each. The total score ranges from 0 to 144. Higher scores indicate greater severity of social anxiety.
Number and percentage of participants who are responders (≥50% improvement from Baseline [Day 1]) based on the LSAS total score | Baseline to Week 8
  The Liebowitz Social Anxiety Scale (LSAS) is a clinician-administered scale that is designed to record the severity of subjective anxiety and avoidance behavior across a range of social interaction and performance situations. The fear and avoidance subscale scores range from 0 to 72 each. The total score ranges from 0 to 144. Higher scores indicate greater severity of social anxiety.
Number and percentage of participants who are remitters based on an LSAS total score of <30 | Baseline to Week 8
  The Liebowitz Social Anxiety Scale (LSAS) is a clinician-administered scale that is designed to record the severity of subjective anxiety and avoidance behavior across a range of social interaction and performance situations. The fear and avoidance subscale scores range from 0 to 72 each. The total score ranges from 0 to 144. Higher scores indicate greater severity of social anxiety.
Change in Hamilton Anxiety Rating Scale (HAM-A) total score | Baseline to Week 8
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale that is designed to rate severity of anxiety. The total score ranges from 0 to 56. Higher scores indicate greater severity of anxiety.
Clinical Global Impression - Severity (CGI-S) score | Baseline to Week 8
  The Clinical Global Impression - Severity (CGI-S) score is rated on a 7-point scale, using a range of responses from 1 (normal, not at all ill) through to 7 (among the most extremely ill patients).
Patient Global Impression - Severity (PGI-S) score | Baseline to Week 8
  The Patient Global Impression - Severity (CGI-S) score is rated on a 7-point scale, using a range of responses from 1 (not present) through to 7 (extremely severe).
Change in Depression Anxiety Stress Scale - 21 items (DASS-21, Stress subscale only) | Baseline to Week 8
  The Depression Anxiety Stress Scale - 21 items (DASS-21), Stress subscale ranges from 0 to 21, with higher scores indicating greater stress severity.
Change in University of California, Los Angeles Loneliness Scale 10-items (UCLA LS 10) score | Baseline to Week 8
  The University of California, Los Angeles Loneliness Scale 10-items (UCLA LS 10) score ranges from 10 to 40, with higher scores indicating greater perceived loneliness.
Change in Pittsburgh Sleep Quality Index (PSQI) global score | Baseline to Week 8
  The Pittsburgh Sleep Quality Index (PSQI) global score ranges from 0 to 21, with higher scores indicating worse sleep quality.
Change in State-Trait Anxiety Inventory (STAI) state | Baseline to Week 8
  The State-Trait Anxiety Inventory (STAI) state score ranges from 20 to 80, with higher scores indicating greater anxiety in the moment.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - SOAR Clinical Study Site, Pheonix, Arizona
  - SOAR Clinical Study Site, Encino, California
  - SOAR Clinical Study Site, Los Angeles, California
  - SOAR Clinical Study Site, Oceanside, California
  - SOAR Clinical Study Site, San Jose, California
  - SOAR Clinical Study Site, Jacksonville, Florida
  - SOAR Clinical Study Site, Tampa, Florida
  - SOAR Clinical Study Site, Boston, Massachusetts
  - SOAR Clinical Study Site, Brooklyn, New York
  - SOAR Clinical Study Site, Memphis, Tennessee
  - SOAR Clinical Study Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: No